CLINICAL TRIAL: NCT01214720
Title: A Randomized, Double-blind Study of the Effect of Avastin Plus Gemcitabine and Erlotinib Compared With Placebo Plus Gemcitabine and Erlotinib on Overall Survival in Patients With Metastatic Pancreatic Cancer
Brief Title: A Study of Avastin (Bevacizumab) Added to a Chemotherapeutic Regimen in Patients With Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO17706
Record Dates: First submitted 2010-10-04; First posted 2010-10-05 (Estimated); Results first posted 2014-08-13 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-07

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Bevacizumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: bevacizumab [Avastin]

INTERVENTIONS:
Drug: bevacizumab [Avastin] — Intervenous repeating dose

SUMMARY:
This study will evaluate efficacy, safety and tolerability of Avastin versus placebo added to a chemotherapeutic regimen in patients with metastatic pancreatic cancer. The anticipated time of study treatment is until confirmed evidence of disease progression, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* metastatic pancreatic cancer (adenocarcinoma);
* good liver, kidney, and bone marrow function.

Exclusion Criteria:

* previous systemic treatment for metastatic pancreatic cancer;
* pregnant or lactating females;
* fertile men, or women of childbearing potential, not using adequate contraception;
* major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start;
* current or recent treatment (within 30 days prior to starting study treatment) with another investigational drug, or participation in another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2005-07; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (90):
- Australia (8):
  - Adelaide
  - Camperdown
  - Footscray
  - Heidelberg
  - Kurralta Park
  - Melbourne
  - St Leonards
  - Sydney
- Austria (4):
  - Graz
  - Innsbruck
  - Salzburg
  - Vienna
- Belgium (4):
  - Antwerp
  - Brussels
  - Leuven
  - Wilrijk
- Canada (6):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Ottawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- China (2):
  - Beijing
  - Shanghai
- Czechia (2):
  - Brno
  - Hradec Králové
- Helsinki, Finland
- France (10):
  - Besançon
  - Bordeaux
  - Boulogne-Billancourt
  - Clichy
  - Limoges
  - Marseille
  - Paris
  - Rouen
  - Saint-Herblain
  - Strasbourg
- Germany (12):
  - Berlin
  - Bochum
  - Bonn
  - Halle
  - Hamburg
  - Heidelberg
  - Leipzig
  - Magdeburg
  - Mainz
  - Mönchengladbach
  - München
  - Trier
- Israel (4):
  - Kfar Saba
  - Petah Tikva
  - Rehovot
  - Tel Aviv
- Italy (9):
  - Bergamo
  - Bologna
  - Brescia
  - Chieti
  - Genova
  - Napoli
  - Orbassano
  - Parma
  - San Giovanni Rotondo
- Amsterdam, Netherlands
- New Zealand (2):
  - Auckland
  - Christchurch
- Lima, Peru
- Poland (4):
  - Gliwice
  - Lublin
  - Szczecin
  - Wroclaw
- Singapore, Singapore
- South Africa (2):
  - Cape Town
  - Pretoria
- Spain (7):
  - Alicante
  - Barcelona
  - Córdoba
  - Elche
  - Madrid
  - Santander
  - Valencia
- Stockholm, Sweden
- Taiwan (2):
  - Kueishan
  - Taipei
- United Kingdom (7):
  - Glasgow
  - Leicester
  - London
  - Manchester
  - Northwood
  - Sutton
  - Truro

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab + Gemcitabine + Erlotinib: Cycle 1 (8-week cycle): Participants received bevacizumab 5 milligrams per kilogram (mg/kg) intravenously (IV) on Days 1, 15, 29, and 43 (followed by 1 week off); gemcitabine 1000 mg per square meter (mg/m^2) IV on Days 1, 8, 15, 22, 29, 36, and 43 (followed by 1 week off); and erlotinib 100 mg tablets/capsules, orally (PO), once daily (QD) for 8 weeks.
  Cycles 2 and beyond (4-week cycle): Participants received bevacizumab 5 mg/kg IV on Days 1 and 15 (followed by 2 weeks off); gemcitabine 1000 mg/m^2 IV on Days 1, 8, and 15 (followed by 1 week off); and erlotinib 100 mg tablets/capsules PO QD. Participants continued on treatment until disease progression, unacceptable toxicity, or participant withdrawal.
- Placebo + Gemcitabine + Erlotinib: Cycle 1 (8-week cycle): Participants received placebo IV on Days 1, 15, 29, and 43 (followed by 1 week off); gemcitabine 1000 mg/m^2 IV on Days 1, 8, 15, 22, 29, 36, and 43 (followed by 1 week off); and erlotinib 100 mg tablets/capsules, PO, QD for 8 weeks.
  Cycles 2 and beyond (4-week cycle): Participants received placebo IV on Days 1 and 15 (followed by 2 weeks off); gemcitabine 1000 mg/m^2 IV on Days 1, 8, and 15 (followed by 1 week off); and erlotinib 100 mg tablets/capsules PO QD. Participants continued on treatment until disease progression, unacceptable toxicity, or participant withdrawal.
Period: Overall Study
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib
Started | 306 | 301
Completed | 221 (Indicates patients who had died at the time of the data cut-off) | 233 (Indicates patients who had died at the time of the data cut-off)
Not Completed | 85 | 68
Not completed — Alive and still on treatment | 34 | 18
Not completed — Alive and in follow-up | 45 | 48
Not completed — Lost to Follow-up | 6 | 2

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All 607 participants randomized to treatment.
Groups:
- Bevacizumab + Gemcitabine + Erlotinib: Cycle 1 (8-week cycle): Participants received bevacizumab 5 mg/kg IV on Days 1, 15, 29, and 43 (followed by 1 week off); gemcitabine 1000 mg/m^2 IV on Days 1, 8, 15, 22, 29, 36, and 43 (followed by 1 week off); and erlotinib 100 mg tablets/capsules, PO, QD for 8 weeks.
  Cycles 2 and beyond (4-week cycle): Participants received bevacizumab 5 mg/kg IV on Days 1 and 15 (followed by 2 weeks off); gemcitabine 1000 mg/m^2 IV on Days 1, 8, and 15 (followed by 1 week off); and erlotinib 100 mg tablets/capsules PO QD. Participants continued on treatment until disease progression, unacceptable toxicity, or participant withdrawal.
- Total: Total of all reporting groups
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib | Total
Number analyzed (Participants) | 306 | 301 | 607
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.5 (10.36) | 61.0 (10.03) | 61.2 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 132 | 113 | 245
  Male | 174 | 188 | 362

OUTCOME MEASURES:

1. Primary Outcome: Duration of Overall Survival - Percentage of Participants With an Event
Description: Duration of overall survival (OS) was defined as the time between date of randomization and date of death due to any cause. Participants without an event were censored at the date last known to be alive. Participants who were randomized but not exposed to study drug and had no further follow up were censored at the date of randomization.
Time Frame: Randomization, Weeks 1-8 of Cycle 1, Weeks 1-3 of consecutive cycles, 28 days and 3 months after lst treatment, and every 3 months for up to 18 months from last participant randomized
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib
Number analyzed (Participants) | 306 | 301
percentage of participants | 72.2 | 77.4

2. Secondary Outcome: Clinical Benefit Response (CBR)
Time Frame: as for outcome 1
Population: The analysis of the CBR was dependent on the calculation of analgesic therapy (AT); this calculation relies on established conversion factors for different morphine derivatives (MD). Many MD utilized by participants do not have well-established conversion factors, yielding uninterpretable results. Therefore, CBR was not analyzed in this study.
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Progression-Free Survival (PFS) - Percentage of Participants With an Event
Description: PFS was defined as the time between the date of randomization and the date of documented progressive disease (PD) defined according to modified Response Evaluation Criteria in Solid Tumors (RECIST) evaluation, or date of death due to any cause. PD was defined as at least a 20 percent (%) increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum (LD) recorded since the treatment started. Participants without an event were censored at the date of last follow up for progression, or date of last available tumor assessment if no further follow up assessment for progression was performed. Participants who were randomized but not exposed to study drug and had no further follow up were censored at the date of randomization.
Time Frame: Screening, Weeks 8, 16, 24, 32, 40, and every 12 weeks thereafter or until confirmed evidence of disease progression
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib
Number analyzed (Participants) | 306 | 301
percentage of participants | 84.0 | 92.4

4. Secondary Outcome: Progression-Free Survival (PFS) - Time to Event
Description: PFS was defined as the time between the date of randomization and the date of documented PD (per RECIST), or date of death due to any cause. Data for participants without an event were censored at the date of last follow up for progression, or date of last available tumor assessment if no further follow up assessment for progression was performed. Participants who were randomized but not exposed to study drug and had no further follow up were censored at the date of randomization. Median PFS was estimated using the Kaplan-Meier method.
Time Frame: Screening, Weeks 8, 16, 24, 32, 40, and every 12 weeks thereafter or until confirmed evidence of disease progression
Population: ITT Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib
Number analyzed (Participants) | 306 | 301
months | 4.6 [3.9 to 5.4] | 3.6 [3.4 to 3.7]
Statistical Analysis 1: Comparison: Bevacizumab + Gemcitabine + Erlotinib vs Placebo + Gemcitabine + Erlotinib; Test type: Superiority or Other; p = 0.0002, Log Rank; Hazard Ratio (HR) = 0.73, 95% CI 2-sided [0.61 to 0.86]

5. Secondary Outcome: Percentage of Participants With Complete Response (CR), Partial Response (PR), or Stable Disease (SD) at First Postbaseline Tumor Assessment
Description: Percentage of participants with CR, PR, or SD according to modified RECIST evaluation at the first postbaseline tumor assessment. CR equaled (=) complete disappearance of all target lesions and non-target disease, with normalization of tumor marker level. PR is greater than or equal to (≥) a 30% decrease of the sum of the LD of all target lesions as referenced to the baseline sum LD of all target lesions. Persistence of one or more non-target lesions(s) and/or maintenance of tumor marker level above normal limits. SD=neither sufficient shrinkage of target lesions to qualify for PR nor sufficient increase to qualify for PD with persistence of one or more non-target lesions(s) and/or maintenance of tumor marker level above normal limits.
Time Frame: Baseline and Week 8
Population: ITT Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib
Number analyzed (Participants) | 306 | 301
percentage of participants | 62.1 [56.4 to 67.6] | 58.5 [52.7 to 64.1]
Statistical Analysis 1: Comparison: Bevacizumab + Gemcitabine + Erlotinib vs Placebo + Gemcitabine + Erlotinib; Test type: Superiority or Other; p = 0.3621, Chi-squared; Approximate 95% confidence interval (CI) for difference of two rates using Hauck-Anderson method; Difference in Response Rates = 3.62, 95% CI 2-sided [-4.3 to 11.6]

6. Primary Outcome: Duration of Overall Survival - Time to Event
Description: Duration of OS was defined as the time between date of randomization and date of death due to any cause. Participants without an event were censored at the date last known to be alive. Participants who were randomized but not exposed to study drug and had no further follow up were censored at the date of randomization. Median duration of survival was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 1
Population: ITT Population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib
Number analyzed (Participants) | 306 | 301
months | 7.1 [6.4 to 7.8] | 6.0 [5.5 to 6.7]
Statistical Analysis 1: Comparison: Bevacizumab + Gemcitabine + Erlotinib vs Placebo + Gemcitabine + Erlotinib; Test type: Superiority or Other; p = 0.2087, Log Rank; Hazard Ratio (HR) = 0.89, 95% CI [0.74 to 1.07]

7. Secondary Outcome: Bevacizumab Concentration in the Presence of Gemcitabine and Erlotinib
Description: Blood samples were collected from a subgroup of participants, in selected centers for the determination of bevacizumab serum concentration before the first bevacizumab/placebo exposure (Week 1) and at Weeks 3, 5, 7, and 9. Each time blood samples were collected just (preferably within 1 hour) before the start of the study treatment.
Time Frame: Weeks 1, 3, 5, 7, and 9
Population: ITT Population. Number (n) = number of participants assessed at a specific visit.
Measure: Geometric Mean (Standard Deviation); unit: micrograms/milliliter
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib
Number analyzed (Participants) | 78
micrograms/milliliter
  Week 1 (n=4) | 0.52 (14.98)
  Week 3 (n=78) | 27.09 (18.23)
  Week 5 (n=73) | 35.23 (24.88)
  Week 7 (n=72) | 41.19 (19.68)
  Week 9 (n=61) | 44.60 (22.57)

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) were reported from Day 1 (or prior to Day 1 for serious AEs [SAEs] related to study specific procedures) until 28 days after last dose. Related nonserious SAEs occurring up to 6 months after last dose of study drug were reported.
Description: Related SAEs: reported indefinitely; related AEs: followed to return to baseline/stabilizing or causal relationship changed. Unrelated, mild/moderate AEs: followed for 28 days after last dose. Severe, life-threatening/related AEs: followed to resolution, causal relationship changed or death.
Arm/Group | Bevacizumab + Gemcitabine + Erlotinib | Placebo + Gemcitabine + Erlotinib
Serious Adverse Events (participants affected / at risk) | 139/297 | 119/286
Other Adverse Events (participants affected / at risk) | 290/297 | 276/286
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Gemcitabine + Erlotinib (N=297) | Placebo + Gemcitabine + Erlotinib (N=286)
Abdominal pain (Gastrointestinal disorders) | 5 | 2
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 2 | 4
Intestinal obstruction (Gastrointestinal disorders) | 3 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 2
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 1
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Ileus paralytic (Gastrointestinal disorders) | 2 | 0
Peritonitis (Gastrointestinal disorders) | 2 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 2
Anal fistula (Gastrointestinal disorders) | 1 | 0
Anal ulcer (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 0 | 1
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1 | 0
Sigmoiditis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 8 | 6
Pneumonia (Infections and infestations) | 9 | 2
Abdominal abscess (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 0 | 3
Septic Shock (Infections and infestations) | 0 | 3
Bacterial sepsis (Infections and infestations) | 2 | 0
Biliary tract infection (Infections and infestations) | 0 | 2
Escherichia sepsis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Subcutaneous abscess (Infections and infestations) | 2 | 0
Abscess (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Biliary sepsis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Central line infection (Infections and infestations) | 0 | 2
Disseminated cytomegaloviral infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Infected insect bite (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 1
Pilonidal cyst (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Pneumonia klebsiella (Infections and infestations) | 0 | 1
Renal cyst infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 12
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pyrexia (General disorders) | 16 | 11
General physical health deterioration (General disorders) | 1 | 3
Asthenia (General disorders) | 1 | 2
Oedema peripheral (General disorders) | 0 | 2
Death (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 5 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Acquired haemophilia with anti FVIII, XI, or XIII (Blood and lymphatic system disorders) | 1 | 0
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 5
Thrombosis (Vascular disorders) | 1 | 2
Aortic dissection (Vascular disorders) | 0 | 1
Cardiovascular insufficiency (Vascular disorders) | 0 | 1
Haemorrhage (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 0 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 4 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 1
Jaundice (Hepatobiliary disorders) | 3 | 0
Biliary dilatation (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Gallbladder perforation (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 2 | 3
Cerebral infarction (Nervous system disorders) | 1 | 1
Syncope (Nervous system disorders) | 1 | 1
Cerebral artery embolism (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 1
Stent occlusion (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatic haematoma (Injury, poisoning and procedural complications) | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Renal impairment (Renal and urinary disorders) | 2 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 2 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
C-reactive protein increased (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Oedema genital (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Ileectomy (Surgical and medical procedures) | 1 | 0
Vomiting (Gastrointestinal disorders) | 8 | 4
Renal failure acute (Renal and urinary disorders) | 0 | 1
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Malabsorption (Gastrointestinal disorders) | 0 | 1
Intra-abdominal haematoma (Gastrointestinal disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Perianal abcess (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Hypercreatinaemia (Musculoskeletal and connective tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab + Gemcitabine + Erlotinib (N=297) | Placebo + Gemcitabine + Erlotinib (N=286)
Diarrhoea (Gastrointestinal disorders) | 145 | 144
Nausea (Gastrointestinal disorders) | 135 | 146
Vomiting (Gastrointestinal disorders) | 108 | 118
Constipation (Gastrointestinal disorders) | 79 | 65
Abdominal pain (Gastrointestinal disorders) | 46 | 39
Abdominal pain upper (Gastrointestinal disorders) | 33 | 29
Stomatitis (Gastrointestinal disorders) | 34 | 19
Dyspepsia (Gastrointestinal disorders) | 25 | 20
Flatulence (Gastrointestinal disorders) | 19 | 10
Fatigue (General disorders) | 104 | 97
Pyrexia (General disorders) | 94 | 99
Oedema peripheral (General disorders) | 51 | 49
Asthenia (General disorders) | 41 | 44
Mucosal inflammation (General disorders) | 25 | 29
Chills (General disorders) | 18 | 15
Rash (Skin and subcutaneous tissue disorders) | 146 | 126
Alopecia (Skin and subcutaneous tissue disorders) | 40 | 44
Dry skin (Skin and subcutaneous tissue disorders) | 37 | 23
Acne (Skin and subcutaneous tissue disorders) | 30 | 17
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 25 | 19
Pruritus (Skin and subcutaneous tissue disorders) | 22 | 18
Anaemia (Blood and lymphatic system disorders) | 77 | 96
Thrombocytopenia (Blood and lymphatic system disorders) | 93 | 76
Neutropenia (Blood and lymphatic system disorders) | 87 | 75
Leukopenia (Blood and lymphatic system disorders) | 16 | 20
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 89 | 32
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 31 | 26
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 24
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Headache (Nervous system disorders) | 39 | 24
Dysgeusia (Nervous system disorders) | 35 | 26
Dizziness (Nervous system disorders) | 20 | 23
Anorexia (Metabolism and nutrition disorders) | 64 | 66
Insomnia (Psychiatric disorders) | 35 | 25
Depression (Psychiatric disorders) | 15 | 18
Anxiety (Psychiatric disorders) | 18 | 10
Hypertension (Vascular disorders) | 58 | 28
Back pain (Musculoskeletal and connective tissue disorders) | 21 | 22
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 9
Urinary tract infection (Infections and infestations) | 29 | 17
Weight decreased (Investigations) | 15 | 21
Proteinuria (Renal and urinary disorders) | 15 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.